CLINICAL TRIAL: NCT01697423
Title: Comparative Assessment of Intra-articular Knee Injections of Platelet-rich Plasma (PRP) and Hyaluronic Acid in the Treatment of Knee Osteoarthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012-003565-18; 2011-25 (Other: AP HM)
Record Dates: First submitted 2012-09-28; First posted 2012-10-02 (Estimated); Last update posted 2023-04-21 (Actual); Status verified 2017-07

CONDITIONS: the Treatment of Knee Osteoarthritis

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- platelet-rich plasma (Experimental)
  Interventions: Drug: platelet-rich plasma
- durolane (Active Comparator)
  Interventions: Drug: durolane

INTERVENTIONS:
Drug: platelet-rich plasma
  Arms: platelet-rich plasma
Drug: durolane
  Arms: durolane

SUMMARY:
The incidence of cartilage pathology has grown due to the ageing population, and the increase in sports participation and its associated trauma. The aim of the treatment of symptomatic osteoarthritis consists in reducing pain and improving the knee function in order to limit the sport, professional and social negative impact in the youngest patients.

The symptomatic treatment of knee osteoarthritis associates painkillers and non steroid anti inflammatory drugs (nsad). In case of ineffectiveness of the oral drugs intra articular injections are proposed.

Intra articular injections of hyaluronic acid are recommended by the American College of Rheumatology and the European League against Rheumatism for the treatment of knee osteoarthritis. Nevertheless their efficacy remain non predictable in patients so as the duration of clinical improvement which does not exceed 6 months.

The articular cartilage has a limited capacity for self-repair due to the low mitotic activity of chondrocytes and its avascularity.

Platelet-rich plasma is a natural concentrate of growth factors: PDGF, TGF b, IGF-1, FGF and the cytokines, liberated by platelet degranulation. The influence of these growth factors in the cartilage repair is being widely investigated in vivo and in vitro. These factors could stimulate the chondral reparation via a neovascularization, a collagen synthesis and an activation of the chondrocytes.

The hypothesis is that the intra articular injection of PRP, with its capacity to enhance articular cartilage repair, could be a therapeutic alternative to hyaluronic acid in the treatment of knee osteoarthritis resisting the oral drugs.

Material and methods: We intend to conduct a comparative, monocentric prospective randomized, double-blind study on 80 patients with symptomatic knee osteoarthritis to compare the results of 2 intra articular treatment: platelet-rich plasma and hyaluronic acid.

ELIGIBILITY:
Inclusion Criteria:

* 1. Males and females between 20 to 75 years of age 2. Symptomatic knee arthritis 3. Axial deformity of the lower limb equal or lower than 5° 4. BMI between 20 to 30 5. Written informed consent, signed by patient or legal representative (if patient unable to sign).

  6. HB > 10g/dl 7. Negative pregnancy test

Exclusion Criteria:

1. Axial deformity of the lower limb over 5°
2. Knee instability
3. BMI < 20 or > 30
4. Thrombocytopenia < 150 G/L
5. Thrombopathy
6. Anaemia: HB < 10g/dl
7. Positive serology VIH1 and 2, Agp24, Ac HCV, Ag HbS, AcHbc, Ac HTLV I and II, TPHA
8. Chronic treatment by corticosteroid per os or treatment completed more than 2 weeks before inclusion
9. Intra articular knee injection of corticosteroid or completed more than 8 weeks before inclusion
10. Intra articular knee injection of hyaluronic or completed more than 24 weeks before inclusion
11. NSAI treatment completed more than 2 weeks before inclusion
12. Fever or recent disease
13. Auto immune disease
14. Inflammatory Arthritis
15. Immune deficit
16. Infectious disease
17. Pregnancy
18. Patient under guardianship.
19. Participation in another investigational trial within this trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Actual)
Dates: Start 2012-12-11 (Actual); Primary Completion 2016-03-30 (Actual); Study Completion 2017-11-29 (Actual)

PRIMARY OUTCOMES:
Variation of the functional score of WOMAC | 12 months
  evaluate the non inferiority between platelet-rich plasma (PRP) and hyaluronic acid. onthé evolution of the knee function, by assessing the difference with a functional score (WOMAC), before and 3 months after treatment.

SECONDARY OUTCOMES:
the evolution of pain | 12month

CONTACTS AND LOCATIONS:
Overall Officials: BERNARD BELAIGUES, Study Director — Assistance Publique Hopitaux De Marseille; marie laure LOUIS, Principal Investigator — AP HM
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France